CLINICAL TRIAL: NCT00634153
Title: The Surgical Gastrointestinal Diseases Registry Protocol
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Randall Brand, Professor of Medicine, University of Pittsburgh
Other Study IDs: 03-145
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Research Registry — We are asking for permission to allow us to place subject's past, current and future medical record information into a Surgical Gastrointestinal Disease Registry. By placing the medical record information of many subjects into a research registry, researchers will be able to conduct research studies directed at increasing our knowledge about Gastrointestinal Diseases.

SUMMARY:
By placing the medical record information of many subjects into a research registry, researchers will be able to conduct research studies directed at increasing our knowledge about Gastrointestinal Diseases.

DETAILED DESCRIPTION:
Researchers are asking for past, current and future medical record information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects being seen by the University of Pittsburgh Medical Center for gastrointestinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2004-01; Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Allow researchers to review and study the medical records of many individuals to answer questions about their disease and its treatment. | 1-N/A

SECONDARY OUTCOMES:
It will help researchers identify and recruit subjects who are eligible for participation in future research studies. | 1-N/A

CONTACTS AND LOCATIONS:
Overall Officials: Randall E. Brand, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States